CLINICAL TRIAL: NCT02534415
Title: Effect of Topically-Applied Hyaluronic-Acid on Palatal Epithelial Wound Closure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YU-351
Record Dates: First submitted 2015-08-17; First posted 2015-08-27 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Wound Healing Complication
Keywords: Antiinflammatory; Gingiva; Hyaluronic acid; Palate; Transplants; Wound healing
MeSH Terms: interventions — Peripac

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Periodontal dressing material (Active Comparator): Palatal wound area was covered with periodontal dressing material at baseline and 3rd day
  Interventions: Drug: Periodontal dressing material
- 0.2% Hyaluronic acid gel (Experimental): 0.2% topical hyaluronic-acid gel was applied to palatal wound area and covered with periodontal dressing material (Peripac®) at baseline and 3rd day
  Interventions: Drug: 0.2% Hyaluronic acid gel
- 0.8% Hyaluronic acid gel (Experimental): 0.8% topical hyaluronic-acid gel was applied palatal wound area and covered with periodontal dressing material (Peripac®) at baseline and 3rd day
  Interventions: Drug: 0.8% Hyaluronic acid gel

INTERVENTIONS:
Drug: Periodontal dressing material — Procedure:Palatal wound area was covered with periodontal dressing material at baseline and 3rd day
  Other Names: Peripac®
  Arms: Periodontal dressing material
Drug: 0.2% Hyaluronic acid gel — 0.2% topical hyaluronic-acid gel was applied to palatal wound area and covered with periodontal dressing material (Peripac®) at baseline and 3rd day
  Other Names: Gengigel
  Arms: 0.2% Hyaluronic acid gel
Drug: 0.8% Hyaluronic acid gel — 0.8% topical hyaluronic-acid gel was applied palatal wound area and covered with periodontal dressing material (Peripac®) at baseline and 3rd day
  Other Names: Gengigel
  Arms: 0.8% Hyaluronic acid gel

SUMMARY:
Aim of the study is to assess the therapeutic effects of topical hyaluronic-acid use on secondary wound healing of the free gingival graft donor site. The hypothesis of this study is that topical hyaluronic-acid gel has positive effects on secondary wound healing of free gingival graft donor site by reducing pain, burning sensation, and accelerating the healing.

DETAILED DESCRIPTION:
The objective of the randomized, single blind, controlled and parallel clinical trial was to assess therapeutic effects of topical hyaluronic-acid on secondary wound healing of free gingival graft donor site.

Primary outcome variables that pain and burning sensation changes were assessed at 3, 7, 14, 21 days after surgery by the examiner. Pain and burning sensation were assessed by patients using the VAS, score 0 indicate no pain or burning sensation, score 10 indicate severe pain or burning sensation. Secondary outcome variables included color match, consistency and epithelization of the wound area. These parameters were assessed by the same examiner at 3, 7, 14, 21 and 42 days after surgery. Color of the palatal mucosa was assessed by comparing it to that of the adjacent and opposite site using the VAS. Score 0 indicate no color match and score 10 indicate very good color match. Consistency of the palatal mucosa was assessed with a blunt instrumentation and scored as soft or firm. Epithelialization was scored clinically as none, partial or complete.

Sample size has been estimated in 12 subjects per treatment groups. Random allocation of the treatment sites to test and control groups will be performed using a computerized selection of random numbers for allocation of the study groups.

Clinical images obtained at baseline, 3, 7, 14, 21 and 42 days after surgery from each treatment site.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* No periodontal surgical treatment in the previous 6 months on the involved sites

Exclusion Criteria:

* Smoking
* Patients with a pregnancy or lactation period
* Self-reported history of antibiotic medication within three months
* Absence of tooth in the area of donor site

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-08; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Pain | 21 days
  Using a visual analog scale (0: No pain, 10: Severe pain)

SECONDARY OUTCOMES:
Color match | 42 days
  Using a visual analog scale (0: No color match, 10: Good color match) (Adjacent and opposite site)
Consistency | 42 days
  Soft/firm
Epithelialisation | 42 days
  None/partial/complete
Burning Sensation | 21 days
  Using a visual analog scale (0: No burning sensation, 10: Severe burning sensation)

CONTACTS AND LOCATIONS:
Overall Officials: Bahar Kuru, Prof. Dr., Study Director — Marmara University, Faculty of Denistry, Department of Periodontology; Başak Doğan, Prof. Dr., Study Chair — Marmara University, Faculty of Denistry, Department of Periodontology; Hatice Selin Yıldırım, Dr., Principal Investigator — Marmara University, Faculty of Denistry, Department of Periodontology